CLINICAL TRIAL: NCT07337213
Title: Knee Extensor-Focused Biomechanical Intervention for Pain, Posture, and Disability in Non-Specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effect of Knee Extensor Training on the Lumbar Spine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lincoln University College (Other)
Collaborators: Cairo University (Other); Taif University (Other)
Responsible Party: Principal Investigator, ALHUMAYANI ABDULLAH FALEHA, Principal investigator, Lincoln University College
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUC/RADMIN/SP/05/903
Record Dates: First submitted 2025-12-09; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Non Specific Low Back Pain
MeSH Terms: interventions — Conization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- control group (Active Comparator): lumbar strengthening
  Interventions: Other: back strengthening exercise
- Treatment Group I (Experimental): lumbar strengthening exercise and knee CKC exercise
  Interventions: Other: OKC Exercise
- Treatment Group II (Experimental): lumbar strengthening exercise and knee CKC exercise
  Interventions: Other: CKC Exercise
- Treatment Group III (Experimental): lumbar strengthening exercise and knee OKC and CKC exercise
  Interventions: Other: CKC and OKC Exercise

INTERVENTIONS:
Other: back strengthening exercise — strengthening exercise to lumbar extensors
  Arms: control group
Other: OKC Exercise — knee extensor OKC exercise added to the lumbar strengthening exercise
  Arms: Treatment Group I
Other: CKC Exercise — knee extensor CKC exercise added to the lumbar strengthening exercise
  Arms: Treatment Group II
Other: CKC and OKC Exercise — knee extensor OKC and CKC exercise added to the lumbar strengthening exercise
  Arms: Treatment Group III

SUMMARY:
The goal of this clinical trial is to learn if knee extensor training with different protocols works to treat LBP in adults.. The main questions it aims to answer are:

What are the comparative effects of open and closed kinetic chain knee extensor strengthening exercises versus lumbar stabilization exercises on lumbar curvature, postural control, and disability in individuals with non-specific low back pain? 1.4.2. How does open kinetic chain knee extensor strengthening affect pain, functional capacity, and lumbar spine stability compared to closed kinetic chain exercises in individuals with non-specific low back pain? 1.4.3 What is the effect of open kinetic chain knee extensor strengthening on pain, functional capacity, and lumbar spine stability compared to conventional lumbar muscle exercises in individuals with non-specific low back pain? 1.4.4 What is the effect of closed kinetic chain knee extensor strengthening on pain, functional capacity, and lumbar spine stability compared to conventional lumbar muscle exercises in individuals with non-specific low back pain? 1.4.5 What is the effect of open kinetic chain knee extensor strengthening on pain, functional capacity, and lumbar spine stability in individuals with non-specific low back pain? 1.4.6 What is the effect of close kinetic chain knee extensor strengthening on pain, functional capacity, and lumbar spine stability in individuals with non-specific low back pain? 1.4.7 What is the effect of conventional lumbar extensor strengthening on pain, functional capacity, and lumbar spine stability in individuals with non-specific low back pain Researchers will compare three different exercise protocols to a control group (will not receive exercise) to see if knee extensor training has an effect on problems associated with LBP.

Participants will:

* Exercise three times per week for 8 weeks
* Be assessed before, 4 weeks after, and 8 weeks after intervention

ELIGIBILITY:
Inclusion Criteria:

I. Males aged 40 to 60 years, II. nonsmokers, III. with normal body mass index IV. of Saudi nationality, V. office workers, VI. suffering from chronic NLBP for 12 weeks or more with a moderate disability according to the Oswestry Disability Index (score of 21 - 40%) moderate activity level according to the Arabic version of the International Physical Activity Questionnaire short form .

Exclusion Criteria:

I. Previous spinal surgery, fracture, deformity, or disease. II. Neurological deficit and Lower limb deformity or fracture, or disease. III. Mental or psychological illness. The Arabic version of the Self-Reporting Questionnaire (SRQ-20) developed by the World Health Organization (WHO) to screen for common mental disorders such as depression and anxiety, uses a cut-off score to distinguish between individuals with and without significant psychological distress. A score of 7 or below is generally considered "normal", indicating no significant psychological distress (Al-Subaie et al., 1998).

IV. Systematic chronic illnesses such as hypertension, cardiac and respiratory disorders, and diabetes mellitus.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only males will be recruited for the study
Enrollment: 128 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in the Lumbar lordosis Cobb angle in degrees measured by X-ray | 8 weeks

SECONDARY OUTCOMES:
Mean change of LBP intensity from the baseline measured by Numeric Pain Rating Scale | 8 weeks
  Minimum Value: 0, which represents "no pain". Maximum Value: 10, which represents "worst imaginable pain," "worst possible pain," or "most intense pain imaginable Higher scores indicate a worse outcome
Mean change in the quality of Life score as measured by the Oswestry Disability Index | 8 weeks
  Minimum Value: 0%, which represents the highest possible level of functioning and independence (no disability).
  Maximum Value: 100%, which represents the lowest possible level of functioning and total dependence
Mean change in the muscle strength measured by the Hand-held dynamometer | 8 weeks
  A higher score indicate improvement
Mean change in the posture control measured by the stare exursion test | 8 weeks
  Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: ABDULLAH F ALHUMAYANI, Principal Investigator — LUC Malaysia

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-11-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT07337213/Prot_SAP_ICF_000.pdf